CLINICAL TRIAL: NCT04245410
Title: Surgical Treatment of Pancreatic Metastases From Renal Cell Carcinoma
Acronym: PANMEKID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Head of Surgery, Clinical Professor, Universidad de Extremadura
Other Study IDs: UE-CHUB 001-2020
Record Dates: First submitted 2020-01-25; First posted 2020-01-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Surgical Procedure; Disease Free Survival; Overall Survival
Keywords: Renal cell carcinoma; Pancreatic metastases; Resection
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients surgically treated of pancreatic metastases from RCC: Patients surgically treated of pancreatic metastases from renal cell carcinoma. Pancreaticoduodenectomy, distal pancreatectomy or total pancreatectomy are included.

SUMMARY:
Pancreatic metastases are a rare entity. In cases of metastatic renal carcinoma (RCC) it can present as isolated pancreatic metastasis, considering the possibility of surgical resection.

Goals:

* Define survival after resection of pancreatic cancer metastases renal in a wide range of our country.
* Identify predictive survival factors

Methods:

Retrospective multicenter study in which cases of pancreatic resection due to renal cancer metastases.

DETAILED DESCRIPTION:
Introduction:

Pancreatic metastases are a rare entity and often synonymous with broader dissemination. However, in cases of metastatic renal carcinoma (RCC) it can present as isolated pancreatic metastasis, considering the possibility of surgical resection. Most of the literature refers to isolated cases or short series, with the Johns Hopkins Hospital series being the largest in a single published center (1,2). In all of them, survival after resection is prolonged.

Recently, due to the results obtained with the tyrosine kinase inhibitor drugs, the value of resection of metastases of RCC origin has been questioned in an Italian multicenter study (3), although other studies consider that resection can improve the prognosis if It is associated with these drugs (4).

Justification:

The existing literature is limited to short series or mostly isolated cases. There are no clear prognostic factors that are limited in most cases to being merely descriptive studies.

Goals:

* Define survival after resection of pancreatic cancer metastases renal in a wide range of our country.
* Identify predictive survival factors that allow establishing Subgroups of patients with the greatest benefit after surgery or, conversely, those who potentially do not benefit from drug treatment.

Method:

Retrospective multicenter study in which cases of pancreatic resection due to renal cancer metastases are collected until December 2019, identified by each of the centers included in the study. A data collection sheet has been designed for each case that will be sent to the participating centers. To know which centers could have performed some pancreatic resection due to renal cancer metastases, an email has been sent to all members of the Spanish association of surgeons and Spanish members of International Hepato-pancreatic and biliary surgery association and this information has been included on their websites. The study variables include those related to demographic data of the patient, with the primary tumor, with the presentation of pancreatic metastasis, pancreas surgery and short-term and long-term postoperative follow-up.

Statistic analysis The data will be analyzed using the IBM SPSS Statistics for Mac version 22.0 program (IBM Corp., Orchard Road Armonk, New York, US). Student's t, Mann Whitney U, Chi-square, or Fisher's test will be used according to the parameters studied. Categorical data will be presented as frequency and percentage. Continuous data will be presented as mean and standard deviation or median and interquartile range depending on the distribution of the data. Subgroups created to compare characteristics and results will be measured using Mann Whitney U, Chi-square or Kruskal Wallis test. A p <0.05 will be considered statistically significant.

Limitations of the study:

The main limitation is the retrospective and multicenter nature that can lead to selection or information bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resecable pancreatic metastases from RCC

Exclusion Criteria:

* Unresecable pancreatic metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated from renal cell carcinoma in the past that have developed pancreatic metastases. They are included in the study after pancreatic resection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 60 months
  Overall survival (months) from surgical resection of pancreatic metastases
Disease free survival | Up to 60 months
  Disease free survival (months) from surgical resection of pancreatic metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Gerardo Blanco-Fernández, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tosoian JJ, Cameron JL, Allaf ME, Hruban RH, Nahime CB, Pawlik TM, Pierorazio PM, Reddy S, Wolfgang CL. Resection of isolated renal cell carcinoma metastases of the pancreas: outcomes from the Johns Hopkins Hospital. J Gastrointest Surg. 2014 Mar;18(3):542-8. doi: 10.1007/s11605-013-2278-2. Epub 2013 Oct 26. PMID 24163138
- [Background] Lee SR, Gemenetzis G, Cooper M, Javed AA, Cameron JL, Wolfgang CL, Eckhauser FE, He J, Weiss MJ. Long-Term Outcomes of 98 Surgically Resected Metastatic Tumors in the Pancreas. Ann Surg Oncol. 2017 Mar;24(3):801-807. doi: 10.1245/s10434-016-5619-z. Epub 2016 Oct 21. PMID 27770346
- [Background] Santoni M, Conti A, Partelli S, Porta C, Sternberg CN, Procopio G, Bracarda S, Basso U, De Giorgi U, Derosa L, Rizzo M, Ortega C, Massari F, Iacovelli R, Milella M, Di Lorenzo G, Buti S, Cerbone L, Burattini L, Montironi R, Santini D, Falconi M, Cascinu S. Surgical resection does not improve survival in patients with renal metastases to the pancreas in the era of tyrosine kinase inhibitors. Ann Surg Oncol. 2015;22(6):2094-100. doi: 10.1245/s10434-014-4256-7. Epub 2014 Dec 4. PMID 25472645
- [Background] Chang YH, Liaw CC, Chuang CK. The role of surgery in renal cell carcinoma with pancreatic metastasis. Biomed J. 2015 Mar-Apr;38(2):173-6. doi: 10.4103/2319-4170.137771. PMID 25179721